CLINICAL TRIAL: NCT00977496
Title: Development of a Probiotic Strategy to Prevent or Eliminate Nasal Colonization With S Aureus
Brief Title: Development of a Probiotic Strategy to Prevent or Eliminate Nasal Colonization With S. Aureus
Status: Withdrawn | Type: Observational
Sponsor: Tufts Medical Center (Other)
Responsible Party: Patricia Hibberd, MD, PhD, Tufts Medical Center
Other Study IDs: 8784
Record Dates: First submitted 2009-09-14; First posted 2009-09-15 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Hemodialysis
Keywords: hemodialysis; microbiota; Staphylococcus aureus
MeSH Terms: conditions — Staphylococcal Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Nasal Swab: New chronic hemodialysis patients with no evidence of nasal carriage of Staphylococcus aureus from Boston Dialysis Center Inc., the outpatient hemodialysis clinic of Tufts Medical Center
  Interventions: Procedure: Nasal Swab

INTERVENTIONS:
Procedure: Nasal Swab — Swabs will be moistened in sterile 0.9% sodium chloride solution and rotated in the anterior vestibule of both nares and processed for S aureus cultures and for bacterial DNA extraction.

SUMMARY:
The goal of this study is characterize the changes in bacterial diversity of the nares of hemodialysis patients. Another goal is to determine when hemodialysis patients become colonized with the bacteria Staphylococcus aureus, as nasal colonization with S. aureus is a major risk factor for invasive infection in hemodialysis patients. Fifteen subjects will be recruited into the study. Nasal swabs will be collected every month for six months or until one month after S. aureus colonization in order to determine any changes in the bacterial communities of the nose. Clinical data will also be collected to evaluate the possible influence of external factors on changes in the microbial communities in the patients' noses. This study will provide preliminary data on whether oral- and/or nasal-administered probiotics can eliminate nasal carriage of S. aureus.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged 18 years or older
* On a stable hemodialysis schedule three times a week at Tufts Medical Center outpatient hemodialysis unit
* Able to speak English, Spanish, Cantonese, or Mandarin (One of these languages is spoken by >95% of our hemodialysis population)
* Provides informed consent to participate in the study
* No plans to be absent from the dialysis unit in the next 6 months
* Willingness to report on adverse events during the study period

Exclusion Criteria:

* Patients in which hemodialysis was indicated for acute renal failure secondary to septic shock, acute tubular necrosis, or other condition which is felt to be temporary or secondary to a life threatening illness or likelihood of hemodialysis for less than 6 months.
* Treatment with systemic anti-staphylococcal antibiotic therapy within 30 days prior to enrollment or planned use of topical mupirocin applied to the nares
* Receiving peritoneal dialysis (concordance between the colonizing and infecting strain is not as high as in the hemodialysis population (105))
* Absolute neutrophil count less than 500/mm3 or anticipated fall in neutrophil count < 500/mm3 (e.g. as a result of recent chemotherapy)
* Bleeding diathesis such as platelets count less than 20 or INR >4 within the last 30 days
* On immunosuppressive therapy
* Anticipated renal transplant during the next 6 months
* Evidence of active bowel leak, acute abdomen or colitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from the Boston Dialysis Center Inc outpatient hemodialysis clinic of Tufts Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-05

PRIMARY OUTCOMES:
To describe the clinical variables that may be associated with the acquisition of S aureus nasal colonization, over a six-month period. | Monthly for 6 months or monthly until 1 month after positive nasal swab for S aureus
To refine and test the feasibility of using non culture-based methods to study the microbial ecology and bacterial diversity of the anterior nares in patients starting hemodialysis using 16sRNA sequence analysis. | Monthly for 6 months or monthly until 1 month after positive nasal swab for S aureus
To explore changes in bacterial diversity in the anterior nares over a six-month period and in conjunction with S aureus colonization. | Monthly for 6 months or monthly until 1 month after positive nasal swab for S aureus

CONTACTS AND LOCATIONS:
Overall Officials: Patricia L Hibberd, MD, PhD, Principal Investigator — Tufts Medical Center